CLINICAL TRIAL: NCT01849003
Title: An Open-label Study to Evaluate the Effect of Single Dose GS-6615 on QT, Safety and Tolerability in Subjects With Long QT-3 Syndrome
Brief Title: Study of the Effect of GS-6615 in Subjects With LQT-3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-279-0110
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Long QT Syndrome
Keywords: Long QT Syndrome; LQTS; Long QT-3 Syndrome; LQT-3; prolonged QT interval; GS-6615; late sodium current inhibitor
MeSH Terms: conditions — Long QT Syndrome | interventions — eleclazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): Participants will receive a single 10 mg dose of GS-6615.
  Interventions: Drug: GS-6615
- Cohort 2 (Experimental): Participants will receive a single 20 mg dose of GS-6615.
  Interventions: Drug: GS-6615
- Cohort 3 (Experimental): Participants will receive a single 30 mg dose of GS-6615.
  Interventions: Drug: GS-6615
- Cohort 4 (Experimental): Participants will receive a single 60 mg dose of GS-6615.
  Interventions: Drug: GS-6615
- Cohort 5 (Experimental): Participants will receive single doses of GS-6615 as follows:
  * Day 1: 20 mg (loading dose)
  * Day 2: 40 mg (loading dose)
  * Days 3-7: 6 mg (maintenance dose) once daily
  If a participant has a QTcF value of ≤ 420 msec on 2 consecutive time points after the 20 mg dose on Day 1, the participant will receive the maintenance dose of 6 mg on Day 2.
  Interventions: Drug: GS-6615
- Cohort 6 (Experimental): Participants will receive single doses of GS-6615 as follows:
  * Day 1: 50 mg (loading dose)
  * Day 2-3: 10 mg once daily
  * Days 4-7: 20 mg once daily
  Interventions: Drug: GS-6615

INTERVENTIONS:
Drug: GS-6615 — GS-6615 tablet(s) administered orally

SUMMARY:
This mechanism of action study is to evaluate the effect of oral GS-6615 on the QTc interval in participants with Long QT-3 syndrome. This study will be performed in six cohorts of participants in a sequential manner, four single-dose cohorts followed by two multiple-dose cohorts. Duration of treatment for the single-dose cohorts and multiple-dose cohorts will be 1 day and 7 days, respectively. Participants will be confined at the study center from check-in until completion of assessments at discharge.

Participants will be continuously monitored using real-time telemetry throughout the in-clinic confinement. Physical examinations including vital signs, laboratory analysis, electrocardiograms (ECGs), Holter recordings and echocardiography (ECHO) will be performed at defined time points throughout the study period. Assessment of adverse events and concomitant medications will continue throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between ages 18-65 years (inclusive) at time of screening
2. Documented LQT-3 genotype with one of the following mutations: delta KPQ, R1623Q, N1325S, E1784K, S1787N, D1790G, G1631D, 1795insD, delF1617, R1644H, L409P, F2004L, I1768V, T1304M, A1330T, or F1596I3.
3. QTc > 480 msec in lead V5 at screening
4. Weight of at least 50 kg with body mass index (BMI) between 18 and 30 kg/m^2 (inclusive)
5. Females of childbearing potential must have a negative serum pregnancy test at screening and check-in
6. Females of childbearing potential must agree to utilize protocol recommended highly effective contraception methods from three weeks prior to the single dose of study drug and for 30 days following the single dose of study drug

   a. Females who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least 3 months prior to study dosing
7. Males must agree to utilize a protocol recommended highly effective method of contraception during heterosexual intercourse throughout the study period and for 90 days following last dose of study drug. Periodic abstinence and withdrawal are not acceptable methods of contraception
8. Males must refrain from sperm donation from Day -2 through completion of the study and continuing for at least 90 days from the date of last dose of study drug
9. Willing and able to comply with the requirements of the protocol and directions from the clinic staff
10. Willing to avoid consumption of grapefruit, grapefruit juice and Seville oranges within 2 weeks prior to the single dose of study drug until discharge from the clinic
11. Willing to avoid consumption of nicotine (including nicotine gum) and alcoholic beverages within 2 weeks prior to the single dose of study drug until discharge from the clinic
12. Understand and willing to sign informed consent

Exclusion Criteria:

1. Ongoing or history of any medical or surgical condition that, in the judgment of the Investigator, might jeopardize the individual's safety or interfere with the absorption, distribution, metabolism or excretion of the study drug
2. History of meningitis or encephalitis, seizures, migraines, tremors, myoclonic jerks, sleep disorder, anxiety, syncope, head injuries or a family history of seizures
3. Any abnormal electrocardiographic (ECG) findings (except QTc > 460 msec) at screening judged to be clinically significant by the investigator
4. Any abnormal laboratory value or physical examination finding at screening or check-in that is judged by the investigator as clinically significant
5. History of positive serology test for HIV, or hepatitis B or C
6. Positive urine drug test for ethanol, barbiturates, cocaine, opiates, or amphetamines at screening or check-in
7. Positive urine cotinine test at check-in
8. Current treatment with drugs affecting the QT interval
9. Current treatment with sodium-channel blockers, eg, flecainide and mexiletine
10. Current treatment with strong or moderate inhibitors or inducers of cytochrome P450 (CYP)3A4 and 1A2
11. Prior treatment with ranolazine within 7 days prior to study drug administration
12. Use of systemic prescription medications or over-the-counter (OTC) medication, including multivitamins, and dietary and herbal supplement within 2 weeks or 5 times the terminal half-lives of the medication (whichever is longer) prior to the single dose of study drug, and for the duration of the study
13. Use of any experimental or investigational drug or device within 30 days prior to the single dose of study drug or 5 half-lives of the drug, whichever is longer
14. Females who are pregnant or lactating
15. History of drug or alcohol abuse within 12 months prior to initial dosing of study drug
16. Psychosocial or addictive disorders that would interfere with ability to give informed consent or could compromise compliance with the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Changes in QTc intervals (Fridericia formula) | Baseline through Day 7
  Changes in QTc intervals (Fridericia formula; QTcF) from the time-matched ECG in the primary lead V5. In case QT cannot be measured in lead V5, lead II will be designated as the primary lead
  * Change from the time-matched ECG on Day -1 to Day 1 for Cohorts 1-4
  * Change from the time-matched ECG average of Day -1 and Day -2 to Days 1-7 for Cohort 5 and 6

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Baseline through Day 22
Changes in ECHO parameters | Baseline through Day 7
  ECHO parameters relevant for measurement of diastolic function will be assessed.
Area under the plasma concentration-time curve (AUC) from time 0 to the last quantifiable concentration of GS-6615 | Baseline through Day 12
Maximum observed plasma concentration (Cmax) of GS-6615 | Baseline through Day 12
Time to maximum observed concentration (Tmax) of GS-6615 | Baseline through Day 12
Changes in ECG parameters | Baseline through Day 12
  ECG parameters assessed will include PR, RR, QRS, and QT.
  * PR: electrocardiographic interval occurring between the onset of the P wave and the QRS complex representing time for atrial and ventricular depolarization, respectively
  * RR: electrocardiographic interval representing the time measurement between the R wave of one heartbeat and the R wave of the preceding heartbeat
  * QRS: electrocardiographic deflection between the beginning of the Q wave and termination of the S wave representing time for ventricular depolarization
  * QT: electrocardiographic interval between the beginning of the Q wave and termination of the T wave representing the time for both ventricular depolarization and repolarization to occur
Changes in QTc interval (Bazett [QTcB]) | Baseline through Day 7
  Changes in QTcB from the time-matched ECG in the primary lead V5. In case QT cannot be measured in lead V5, lead II will be designated as the primary lead
  * Change from the time-matched ECG on Day -1 to Day 1 for Cohorts 1-4
  * Change from the time-matched ECG average of Day -1 and Day -2 to Days 1-7 for Cohort 5 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Layug, MD, Study Director — Gilead Sciences
Locations (1):
- University of Rochester Medical Center/Strong Memorial Hospital, Rochester, New York, United States